CLINICAL TRIAL: NCT06125808
Title: A Phase 2B, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-finding, Efficacy and Safety Study of HRO350 in Patients with Mild-to-moderate Psoriasis (the 'HeROPA' Study).
Brief Title: Efficacy and Safety Study of HRO350 in Patients with Mild-to-moderate Psoriasis (the 'HeROPA' Study).
Acronym: HeROPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arctic Bioscience (Industry)
Collaborators: Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRO350-PS-2B 'HeROPA'; 2021-003684-96 (EudraCT Number)
Record Dates: First submitted 2023-09-08; First posted 2023-11-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1050 mg HRO350 (Experimental): 1050 mg HRO350 daily given as 3 capsules of HRO350 (350 mg) in the morning and 3 capsules of placebo in the evening. Total of 6 capsules daily.
  Interventions: Drug: HRO350; Drug: Placebo
- 2100 mg HRO350 (Experimental): 2100 mg HRO350 daily given as 3 capsules of HRO350 in the morning and 3 capsules of HRO350 in the evening. Total of 6 capsules daily.
  Interventions: Drug: HRO350
- Placebo (Placebo Comparator): Placebo given as 3 capsules of placebo in the morning and 3 capsules of placebo in the evening, Total of 6 capsules daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRO350 — Active substance phospholipid esters from herring roe oil (PEHeRo)
  Arms: 1050 mg HRO350; 2100 mg HRO350
Drug: Placebo — Placebo; as a sunflower oil in capsules similar to the interventional drug product HRO350 in terms of appearance, smell and taste.
  Arms: 1050 mg HRO350; Placebo

SUMMARY:
HRO350 contains an oil-based extract from herring roe (Clupea harengus) in soft capsules and contains phospholipids (complex lipids) which are naturally rich in marine polyunsaturated fatty acids. All the lipids in HRO350 are natural components of the human diet. It is not fully known how HRO350 exerts its effects, however there are indications that it might have a modulatory effect on the inflammatory processes involved in causing psoriasis. The study is a randomised, double-blind, placebo controlled, dose finding, multi-centre, phase 2B study. Approximately 519 patients will be participating in the UK, Norway, Germany, Finland and Poland. Patients will receive either 1050mg or 2100mg HRO0350 daily, or placebo for up to 52 weeks and will be followed up for a further 8 weeks.

DETAILED DESCRIPTION:
This study is a phase 2 multi-national (Norway, Germany, Finland, Poland and the UK), multi-centre (approx 66 sites), randomised, and placebo-controlled study assessing the dose, efficacy and safety of HRO350 in patients with mild-to-moderate psoriasis.

HRO350 contains phospholipids (complex lipids) which are naturally rich in marine polyunsaturated fatty acids that come from herring roe. All the lipids in HRO350 are natural components of the human diet. It is not fully known how HRO350 exerts its effects, however there are indications that it might have a modulatory effect on the inflammatory processes involved in causing psoriasis. There are limited treatment options available for patients with mild-to-moderate psoriasis that provide treatment satisfaction and an improvement in quality of life.

Therefore, the purpose of this study is to investigate the efficacy and safety of HRO350 in patients with mild to moderate psoriasis and help decide which doses should be included for further testing to provide the 'best' or optimal effects of HR0350.

Approximately 519 patients with mild-to-moderate psoriasis will be included in this study. The screening visit will include a review of the eligibility for the study, a physical examination, review of vital signs and blood and urine samples collected as part of the safety assessment along with assessment of their psoriasis severity.

Daily treatment will begin with 3 capsules of either HRO350 or placebo taken in the morning and 3 capsules of either HRO350 or placebo taken in the evening for up to 52 weeks. The patients will be asked to attend the clinic for a total of 8 visits and will receive 8 phone calls for safety checks and assessment of psoriasis severity. The total length of participation will be up to 60 weeks including an 8 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent.
2. Males or females ≥18 years of age.
3. Diagnosis of chronic, active plaque psoriasis of mild to moderate severity since at least 6 months prior to screening.
4. Psoriasis Area and Severity Index (PASI) score ≥ 3 and ≤ 10 at screening and baseline
5. Body Surface Area (BSA) ≥ 3 at screening and baseline
6. Static Physician's Global Assessment (sPGA) ≥ 2 and ≤ 4 at screening and baseline.
7. Males, and females of child-bearing potential1, must be willing to use highly effective methods of birth control during the study period and until 30 days after end of treatment. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:

   * Combined (oestrogen and progestogen containing hormonal contraception associated with inhibition of ovulation -oral

     -intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation -oral

     * injectable
     * implantable
   * intrauterine device
   * intrauterine hormone-releasing system
   * bilateral tubal occlusion
   * vasectomized partner
   * sexual abstinence (if this is the preferred and usual lifestyle of the patient)

     1. Female patients will be considered to be of childbearing potential as per the Clinical Trial Facilitation Group (CTFG) definition of woman of childbearing potential: Fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement is required.

Exclusion Criteria:

1. Diagnosis of other psoriasis clinical subtypes such as guttate, erythrodermic or pustular psoriasis.
2. Phototherapy [(i.e., ultraviolet radiation (UVB), psoralens and long-wave ultraviolet radiation (PUVA)] within 8 weeks of randomisation and during the trial.
3. Any investigational drug administered within 4 weeks of randomisation or <5 times half-lives, whichever is the longer, and during the trial.
4. Systemic anti-psoriatic treatment last 3 months (for biologics last 6 months) before randomisation or during the trial.
5. Topical anti-psoriatic treatment last 2 weeks before randomisation.
6. Any change in anti-inflammatory medication (for other chronic diseases than psoriasis) last 4 weeks before randomisation and during the trial.
7. Any intake of omega-3 fatty acid supplements or medicines last 2 weeks before randomisation and during the trial.
8. Known fish or vegetable oil (including soy) allergy, or allergy to other ingredients in the study medication, placebo or rescue medication.
9. Baseline white blood cell count <3.0x109/L or lymphocyte count <1.0x109/L, or other pathological results identified during a complete blood count, which in the opinion of the investigator may preclude the patient being enrolled.
10. Previous malignancies (except for non-melanoma skin cancer).
11. Symptomatic coronary or cerebral vascular disease.
12. Known congestive heart failure Grade IV by the New York Heart Association
13. Myocardial infarction within 6 months prior to signing the ICF
14. Onset of unstable angina within 6 months prior to signing the ICF
15. Chronic kidney disease as evidenced by a calculated glomerular filtration rate (GFR) < 60ml/min/1.73m2 at screening.
16. Abnormal liver function tests defined by:

a. AST (SGOT), ALT (SGPT) or alkaline phosphatase (ALP) >3x the upper limit of the normal range (ULN). Elevated gamma-GT (GGT) values exceeding >3x ULN are allowed but these GGT cases will be carefully assessed alongside other clinical and laboratory data by the investigator. q. History of severe gastrointestinal problems. r. Ongoing, active infectious disease. s. Known human immunodeficiency virus (HIV)-positive status or suffering from any other immunosuppressive disease. t. History of major psychiatric illness that could interfere with the conduct of the study.

u. Patients with documented or suspected, clinically significant, alcohol (i.e., > 12g/d for women and 24 g/d for men) or drug abuse within the past 12 months.

v. Any other significant, unstable medical condition that would interfere with the completion of the study or interpretation of results.

w. Women of child-bearing potential* must have a negative serum pregnancy test at Visit 1 (Screening) and a negative urine pregnancy test at Visit 2 (Baseline). x. Females who are pregnant, breast feeding, refuse to use birth control methods or who wish to become pregnant during the study period.

y. Unable to comply with the requirements of the study or who in the opinion of the investigator is unable to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with ≥50% reduction in Psoriasis Area and Severity Index (PASI50). | From Baseline to Week 26
  The PASI assesses efficacy in moderate-to-severe psoriasis and quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percentage of body surface area (BSA)" affected. To be included on the study, patients Psoriasis Area and Severity Index (PASI) score needs to be ≥ 3 and ≤ 10, indicating mild-to-moderate Psoriasis.
  The proportion of patients with ≥50% reduction in Psoriasis Area and Severity Index (PASI) from baseline to week 26 will be compared between: HRO350 2100 mg and placebo, and HRO350 1050 mg and placebo.

SECONDARY OUTCOMES:
Comparisons of Psoriasis Area and Severity Index (PASI) scores | From baseline to week 4, 12, 26, 39, 52 and 60
  Comparing proportions of patients with PASI50 from baseline to Week 4, 12, 39, 52 and 60. Comparing proportions of patients with PASI75 from baseline to Week 4, 12, 26, 39, 52 and 60.
  The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of Psoriasis.
Body Surface Area (BSA) | From baseline to week 12, 26, 39, 52 and 60
  The BSA is a measurement of involved skin over the whole body. Assessment of BSA with psoriasis will be estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represents approximately 1% of the total BSA. The surface area of the whole body is made up of approximately 100 palms or "handprints" (each entire palmar surface or "handprint" equates to approximately 1% of total body surface area). A negative change from baseline indicates a reduction of affected BSA.
  The study will look at: percentage of participants with a ≥ 75 percent (%) improvement from baseline in affected BSA (at Week 12, 26, 39, 52 and 60), percent change from baseline in total BSA with psoriasis (at Week 12, 26, 39, 52 and 60), and percentage of participants who achieved BSA ≤ 3% for participants with baseline affected BSA >3% (at Week 12, 26, 39, 52 and 60).
static Physician Global Assessment (sPGA) | Baseline, Week 4, Week 12, Week 26, Week 39, Week 52, and Week 60.
  The static Physician's Global Assessment (sPGA) will be scored periodically to confirm the severity of psoriasis and to assess efficacy of HRO350/placebo. sPGA is an average assessment of all psoriatic lesions, based on erythema, scaling and induration. The total score will be calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). An sPGA response is defined as sPGA score of clear (0) or almost clear (1).
  The study will look at: percentage of Participants with sPGA Score of 'Clear' or 'Almost Clear' (at week 4, 12, 26, 39, 52 and 60), percentage of Participants with sPGA Score 0, 1, 2, 3 and 4, respectively, percentage of Participants with static Physician Global Assessment (sPGA) of Psoriasis Score of 'Clear' or 'Almost Clear' and with at least a 2-point reduction from baseline at Week 12, 26, 39, 52 and 60.
static Physician's Global Assessment (sPGA) x Body Surface Area (BSA) product | From baseline to week 4, 12, 26, 39, 52 and 60
  The product of sPGA and BSA (sPGAxBSA) has been suggested by several groups as an alternative to PASI in this patient group as it accounts for both extent and severity of psoriasis providing an accurate global assessment of disease. The sPGAxBSA score will be calculated by multiplying the static PGA score by the BSA; i.e. with a range from 0 to 400, as the maximum sPGA = 4, and the maximum BSA = 10.
  The study will look at mean change from baseline in sPGAxBSA score at Week 4, 12, 26, 39, 52 and 60.
Scalp PGA (ScPGA) | From baseline to week 4, 12, 26, 39, 52 and 60
  For patients whose psoriasis involves the scale the ScPGA will be employed. The ScPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an Investigator's assessment of the severity of the three primary signs of the disease: erythema, scaling, and induration of the overall scalp. An ScPGA response is defined as an ScPGA score clear (0) or almost clear (1) with at least a 2-point reduction from baseline among participants with a baseline ScPGA score ≥ 2.
  The study will look at percentage of Participants with a Scalp Physician Global Assessment (ScPGA) Response at Week 4, 12, 26, 39, 52 and 60 among Participants with Baseline ScPGA Score ≥ 2.
Use of Rescue Medication | From baseline to week 4, 12, 26, 39, 52 and 60
  Each patient will have available standardised rescue medication for use if the symptoms of psoriasis are not adequately managed by the study medication (HRO350/placebo). Rescue medication in this study is betamethasone valerate 0.1% w/w ointment and may be used for the relief of inflammatory and pruritic manifestations of the psoriasis on an ad hoc basis. Each patient will be dispensed betamethasone valerate at the study start.
  At the end of the study, all returned rescue medication will be weighed. The use of rescue medication will be calculated. The study will look at mean use of rescue medication (measured as grams used) during study; from baseline to end-of-treatment. And, mean number of days, from baseline to end-of-treatment, rescue medication was used; absolute and proportion of days.
SF-36 | Baseline, Week 26 and Week 52
  36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects are summarized as physical and mental health summary scores. The score range for the physical and mental health scores is 0-100 (100=highest level of functioning).
  The study will look at mean change from baseline for the Physical Component in SF-36 at Week 26 and 52, and mean change from baseline for the Mental Component in SF-36 at Week 26 and 52.
Dermatology Life Quality Index (DLQI) | From baseline to week 4, 12, 26, 39, 52 and 60
  The DLQI (Finlay and Khan, 1994) is a self-administered general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). It is calculated by summing the score for each question, resulting in a total score ranging from a maximum of 30 to a minimum of 0 with 30 corresponding to the worst health-related quality of life, and 0 corresponding to the best score. The minimum clinically important difference (MCID) between scores for the DLQI has been defined as a score difference of 4 (Basra et al., 2015).
  The study will look at: DLQI Total Score, mean change from baseline in DLQI Total Score, proportion of patients who achieve a ≥4-point reduction in DLQI, and mean change from baseline in DLQI for each of 10 items at Week 4, 12, 26, 39, 52 and 60.
PSI | From baseline to week 4, 12, 26, 39, 52 and 60
  The Psoriasis Symptom Inventory (PSI) is a validated patient-reported outcome measure assessing patients' perception of 8 different psoriasis signs and symptoms: itch, redness, scaling, burning, stinging, cracking, flaking and pain (Martin et al., 2013; Bushnell et al., 2013; Revicki et al., 2014). Patients will assess the severity of each item on a 5-point Likert-type rating scale from 0 ('not at all') to 4 ('very severe'). The scores for all 8 items are then summed to give a total score with a range of 0-32. In this study, it is the 7-day recall version of the PSI that will be used.
  The study will look at mean change from baseline in PSI Total Score, and mean change from baseline in PSI for each of 8 items at Week 4, 12, 26, 39, 52 and 60.
Patients overall treatment satisfaction | From baseline to week 4, 12, 26, 39, 52 and 60
  The patient's overall satisfaction to treatment of their psoriasis will be assessed at screening and every 3 months using a simple one-dimensional 5-point Likert scale in which the patient will be questioned: 'How satisfied are you with your current treatment for psoriasis today?', and will be asked to rate their satisfaction by a choice between the categories:
  1. very dissatisfied
  2. dissatisfied
  3. neither satisfied nor dissatisfied
  4. satisfied
  5. very satisfied The study will look at mean change from screening in the treatment satisfaction score at Week 12, 26, 39, 52 and 60.
Discontinuation rate | From baseline to week 4, 12, 26, 39, 52 and 60
  The number and rate of patients discontinuing from the study prior to planned completion (i.e., not completing the 52 weeks of treatment and the 8 weeks follow-up period) will be presented, categorized by reasons for discontinuation as an indirect measure of efficacy.
Safety - Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From screening to week 60
  Frequency tables of all safety variables will be analysed and will i.a. include:
  * Frequency of any Treatment-emergent Adverse Events (TEAEs) and SAEs.
  * Frequency of any TEAE by system organ class (SOC), preferred term (PT), severity and relationship of TEAEs to investigational medicinal product.
  * Discontinuation rate: any or due to TEAEs.
  * Frequency of each safety laboratory variable categorised as
    * Below normal range (clinically significant)
    * Below normal range (not clinically significant)
    * Within normal range
    * Above normal range (not clinically significant)
    * Above normal range (clinically significant)
  Further, full narratives of any SAEs will be described in the study report.

CONTACTS AND LOCATIONS:
Locations (49):
- Finland (2):
  - CRST Helsinki Oy, Helsinki
  - CRST Turku Oy, Turku
- Germany (15):
  - Fachklinik, Bad Bentheim
  - Hautmedizin Bad Soden Studienzentrum GmbH, Bad Soden
  - Hautarztpraxis Dr Wildfeuer, Berlin
  - Isa Research - Interdisciplinary Study Organisation, Berlin
  - Universitätsklinikum Dresden Klinik und Poliklinik für Dermatologie, Dresden
  - Proderma, Institut für klinische Studien und innovative Dermatologie, Dülmen
  - Universitätsklinikum Essen, Essen
  - Derma-Study-Centre, Friedrichshafen
  - Universitätsklinikum Heidelberg, Heidelberg
  - University Clinic UKSH Kiel, Kiel
  - Klinikum der Universität München, Munich
  - Universitätsklinikum Münster, Münster
  - Dermatologisches Studienzentrum Hunsrück am Haut -und Laserzentrum, Simmern
  - Hautarztpraxis Dr. Leitz - Studienzentrum Triderm, Stuttgart
  - Hautarztpraxis Dr. med. Matthias Hoffmann, Witten
- Norway (2):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Haukeland
- Poland (4):
  - Centrum Medyczne All-Med, Krakow
  - KO-MED Centra Medyczne, Puławy
  - MICS Centrum Medyczne, Torun
  - Narodowy Instytut Geriatrii, Warsaw
- United Kingdom (26):
  - The Practice of Health, Barry
  - Heart of Bath Medical Partnership, Bath
  - Waterloo Medical Centre, Blackpool
  - St Luke's Hospital, Bradford
  - Concord Medical Centre, Bristol
  - Royal Primary Care Ashgate, Chesterfield
  - Hathaway Medical Centre, Chippenham
  - Rowden Surgery, Chippenham
  - Lakeside Healthcare Research, Corby
  - University Hospital of North Durham, Durham
  - Haven Health, Felixstowe
  - Honiton Surgery, Honiton
  - Oak Tree Surgery, Liskeard
  - Babylon Healthcare GP at Hand, London
  - Luton and Dunstable University Hospital, Luton
  - Kiltearn Medical Centre, Nantwich
  - Newquay Health Centre, Newquay
  - St Clare Medical Centre, Penzance
  - University Hospitals Dorset, Poole
  - Clarence House Medical Centre, Rhyl
  - Sherbourne Medical Practice, Royal Leamington Spa
  - Salford Royal Hospital, Salford
  - Kings Mill Hospital, Sutton in Ashfield
  - Grove Surgery, Thetford
  - Trowbridge Health Centre, Trowbridge
  - West Walk Surgery, Yate